CLINICAL TRIAL: NCT05886374
Title: A Multicenter, Open-Label Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-415S1 in Patients With Advanced Malignant Solid Tumor
Brief Title: A Study of HMPL-415S1 in Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-415-00CH1
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-415S1 (Experimental): HMPL-415S1 will be administered orally once daily in 28 days treatment cycles
  Interventions: Drug: HMPL-415S1

INTERVENTIONS:
Drug: HMPL-415S1 — HMPL-415S1 will be supplied as 0.5 mg, 5 mg and 25 mg capsules

SUMMARY:
The objective of this study is to evaluate the safety, tolerability and PK profile of HMPL-415S1 and determine MTD and/or RP2D in patients with advanced malignant solid tumor.

DETAILED DESCRIPTION:
This study is expected to enroll 36-81 patients, including 26-66 patients for dose escalation, additional 10-15 patients will be enrolled at the dose level of determined RP2D.

ELIGIBILITY:
Inclusion Criteria:

All the following conditions must be met for enrollment:

1. Fully understand this study and voluntarily sign the ICF;
2. Dose escalation Patients with advanced malignant solid tumor confirmed by histopathology or cytology, who have failed, been intolerant or unavailable to, or have none standard treatment for various reasons; Dose expansion phase: Patients with advanced malignant solid tumor confirmed by histopathology or cytology, who have failed, been intolerant or unavailable to, or have none standard treatment for various reasons, carrying aberrant activating mutations in the KRAS pathway；
3. Presence of at least one measurable lesion (RECIST 1.1 criteria);
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 point;
5. Life expectancy ≥ 12 weeks as judged by the investigator;
6. Male of childbearing potential and their heterosexual partners of childbearing potential must agree to use effective methods of contraception.

Exclusion Criteria:

A patient may not participate in this study if any of the following conditions apply:

1. Patients who priorly received SHP2 inhibitors;
2. Receiving the approved systemic antitumor treatment within 4 weeks prior to the first dose, including: chemotreatment, targeted treatment, immunization treatment, biological treatment, etc. (wash-out for 2 weeks for hormone treatment or traditional chinese medicine and chinese patent medicine with clear antitumor indications);
3. Have been in the treatment period of other interventional clinical studies (including small molecule chemicals and large molecule antibodies) within 4 weeks prior to the first dose. If participating in a non-interventional clinical study (eg, epidemiological study), you can enroll in this study; if already in the survival follow-up period of an interventional clinical study, you can enroll in this study.
4. Major surgery or radical radiotreatment (except palliative radiotreatment for metastases to bone lesions) within 4 weeks prior to first dose.
5. Central nervous system (CNS) malignant tumor or known CNS metastasis;
6. Having multiple factors that affect the absorption, distribution, metabolism or excretion of orally administered drugs (such as inability to swallow drugs, frequent vomiting, chronic diarrhoea, etc.);
7. Any other disease, metabolic abnormality, physical examination abnormal, or clinically significant laboratory test abnormality that, in the judgment of the investigator, would compromise patient compliance or give reason to suspect that the patient has a disease or condition that would compromise the interpretation of study results or place the patient at high risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and determine the maximum tolerated dose (MTD) and/or RP2D of HMPL-415S1 as a single oral agent in advanced malignant solid tumor | from Cycle 0Day1 up to Cycle1Day28 (each cycle is 28 days).
  Occurrence of Dose Limiting Toxicities (DLTs) During the DLT Observation Period

SECONDARY OUTCOMES:
To investigate the pharmacokinetic (PK) profile of oral HMPL-415S1 | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days).
  Plasma peak concentration of HMPL-415S1 (Cmax).
AUCinf (Cycle 0 ) of HMPL-415S1 | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days).
  AUCinf: area under the concentration vs. time curve from zero to infinity after single (first)dose.
AUC(0-tlast) (Cycle 0 ) of HMPL-415S1 | from pre-dose to day 5 of cycle 0. (cycle 0 contains 5 days).
  AUC from time zero to the last data point.
Objective Response Rate (ORR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  Percentage of patients with Complete Response(CR) or Partial Response(PR) as the best response evaluated in accordance with RECIST 1.1.
Disease control rate (DCR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  the proportion of patients with CR or PR or stable disease (SD) as the best response, and the duration of SD needs to be ≥6 weeks.
uration of response (DoR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  as the time from the first appearance of CR or PR to PD or death for any reason (whichever comes first), in the patients with objective response.
Time to response (TTR) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  the time from the first dose of HMPL-415S1 to the first objective response.
Progression-free survival (PFS) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  time from the first dose of study treatment to PD or death for any reason, whichever comes first.
Overall survival (OS) | From baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 3 years).
  time from the first dose of study treatment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Yang, Study Director — Hutchison Medipharma Limited
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No